CLINICAL TRIAL: NCT02408913
Title: VRC 208: Phase 1/1b Open-Label Clinical Trial to Evaluate Dose, Safety and Immunogenicity of Recombinant Modified Vaccinia Virus Ankara Ebola Vaccine,VRC-EBOMVA079-00-VP, Administered Alone or as Boost to cAd3-Ebola Vaccines in Healthy Adults
Brief Title: VRC 208: Dose, Safety and Immunogenicity of a Recombinant Modified Vaccinia Virus Ankara Ebola Vaccine, VRC-EBOMVA079-00-VP (MVA-EbolaZ), Administered Alone or as a Boost to cAd3-Ebola Vaccines in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 150107; 15-I-0107
Record Dates: First submitted 2015-04-03; First posted 2015-04-06 (Estimated); Last update posted 2019-04-11 (Actual); Status verified 2017-04-06

CONDITIONS: Healthy Adult Immune Responses to Vaccine
Keywords: Immunity; Ebola Virus; Ebola Hemorrhagic Fever; Healthy; Filovirus
MeSH Terms: conditions — Hemorrhagic Fever, Ebola

ARMS (4):
- Group 2 (Experimental): MVA-EbolaZ 1x10(8) PFU
  Interventions: Biological: VRC-EBOMVA079-00-VP (MVA-EbolaZ)
- Group 3 (Experimental): cAd3-EBO 2x10(11) PU followed by MVAEbolaZ 1x10(8) PFU at 8 weeks
  Interventions: Biological: VRC-EBOMVA079-00-VP (MVA-EbolaZ); Biological: VRC-EBOADC069-00-VP (cAd3-EBO)
- Group1 (Experimental): MVA-EbolaZ 1x10(7) PFU
  Interventions: Biological: VRC-EBOMVA079-00-VP (MVA-EbolaZ)
- Groups 4 to 7 (Experimental): MVA-EbolaZ 1x10(8) PFU administered in VRC 208 to participants who received cAd3-EBO or cAd3-EBOZ in VRC 207.
  Interventions: Biological: VRC-EBOMVA079-00-VP (MVA-EbolaZ)

INTERVENTIONS:
Biological: VRC-EBOMVA079-00-VP (MVA-EbolaZ) — Ebola Modified Vaccinia Virus Ankara Vaccine
Biological: VRC-EBOADC069-00-VP (cAd3-EBO) — Ebola Chimpanzee Adenovirus Vector Vaccine
  Arms: Group 3

SUMMARY:
Background:

- Ebola virus is a rare disease that starts with fever and muscle aches, but can lead to death. The 2014 Ebola outbreak in West Africa is the largest to date. There are no approved treatments for Ebola. Researchers want to see if two new vaccines VRC-EBOMVA079-00-VP (MVA-EbolaZ) and VRC-EBOADC069-00VP ( cAd3-EBO ) are safe and able to induce an immune response against Ebola.

Objectives:

- To see if the two new vaccines are safe and if they cause any side effects. Also, to study immune responses to the vaccines.

Eligibility:

- Healthy adults ages 18-66

Design:

* Participants will get one or two study vaccine injections depending on the study group they are assigned to. Each injection will repeat the same schedule:
* A needle and syringe will inject the vaccine into an upper arm muscle.
* 1-2 days later, participants must call the clinic to report how they feel.
* For 7 days they will check their temperature with a thermometer given to them. They will look at the injection site, and measure any redness or swelling with a ruler. They will write down any symptoms they have.
* In the first 2 months, participants will have at least 6 clinic visits and 1 phone contact. At each visit, participants will be checked for health changes or problems. They will tell how they feel and if they have taken any medications. Blood and urine samples may be collected.
* Participants might need to have extra clinic visits and laboratory tests if they have health changes that need to be checked.

DETAILED DESCRIPTION:
This Phase 1/1b study will examine dose, safety, tolerability and immunogenicity of an investigational MVA-vectored Ebola vaccine in healthy adults. The vaccine encodes wild type (WT) glycoprotein (GP) from Zaire strain of Ebola and will be administered intramuscularly (IM) with needle and syringe. The safety and tolerability of the MVA-EbolaZ will be evaluated at escalating doses of 1x10(7) and 1x10(8) plaque forming units (PFU). Part 1 includes enrollment of vaccine-naive subjects to conduct a dose escalation of the MVA-EbolaZ vaccine and to evaluate the vaccine as a boost for the cAd3-EBO vaccine. In Part 2 of the study, up to 140 subjects who received the cAd3-EBO or cAd3-EBOZ vaccine in VRC 207 study will be boosted with MVA-EbolaZ. The hypotheses are that the study vaccines will be safe and elicit immune responses to Ebola GP, and that the prime-boost regimens will be safe and result in a more polyfunctional response to Ebola GP that is of greater magnitude and duration than response to either of the vaccines alone.

ELIGIBILITY:
* INCLUSION CRITERIA:

Inclusion Criteria for Groups 1, 2, and 3.

A volunteer must meet all of the following criteria to be eligible:

1. 18 to 50 years old.
2. Available for clinical follow-up through the last study visit.
3. Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process.
4. Able and willing to complete the informed consent process.
5. Willing to donate blood for sample storage to be used for future research.
6. In good general health without clinically significant medical history.
7. Physical examination and laboratory results without clinically significant findings and a body mass index (BMI) less than or equal to 40 within the 56 days prior to enrollment.

   Laboratory Criteria within 56 days prior to enrollment:
8. Hemoglobin within institutional normal range or accompanied by the Principal Investigator (PI) or designee approval.
9. White blood cells (WBC) = 3,300-12,000 cells/mm(3).
10. WBC differential either within institutional normal range or accompanied by the PI or designee approval.
11. Total lymphocyte count greater than or equal to 800 cells/mm(3).
12. Platelets = 125,000-400,000/mm(3).
13. Alanine aminotransferase (ALT) less than or equal to 1.25 times upper limit of normal.
14. Serum creatinine less than or equal to 1.1 times upper limit of normal.
15. Partial thromboplastin time (PTT) less than or equal to 1.1 times upper limit of normal or accompanied by the Principal Investigator (PI) or designee approval.
16. Prothrombin time (PT) less than or equal to1.1 times upper limit of normal or accompanied by the Principal Investigator (PI) or designee approval.
17. HIV-uninfected as evidenced by a negative FDA-approved HIV diagnostic blood test.

    -Female-Specific Criteria:
18. Negative beta-HCG (human chorionic gonadotropin) pregnancy test (urine or serum) on day of enrollment if woman is presumed to be of reproductive potential.
19. Agrees to use an effective means of birth control from at least 21 days prior to enrollment through 24 weeks after last study vaccination if presumed to be of reproductive potential.

EXCLUSION CRITERIA:

Exclusion Criteria for Groups 1, 2, and 3

A volunteer will be excluded if one or more of the following conditions apply:

Volunteer has received any of the following substances:

1. Investigational Marburg vaccine in a prior clinical trial.
2. Investigational Ebola vaccine in a prior clinical trial.
3. Investigational cAd3 or MVA vaccines in a prior clinical trial.
4. Evidence of increased cardiovascular disease risk defined as >10% five year risk by the non-laboratory method.
5. Electrocardiogram (ECG) with clinically significant abnormalities (examples may include: pathologic Q waves, significant ST-T wave changes, left ventricular hypertrophy, any non-sinus rhythm excluding isolated premature atrial contractions, right or left bundle branch block, advanced A-V heart block). ECG abnormalities determined by a cardiologist to be clinically insignificant as related to study participation do not preclude study enrollment.
6. Type 1 hypersensitivity reaction to aminoglycoside antibiotics.
7. More than 10 days of systemic immunosuppressive medications except for short-term treatments of minor ailments in otherwise healthy volunteers, or cytotoxic medications within the 4 weeks prior to enrollment, or any within the 14 days prior to enrollment.
8. Blood products within 112 days (16 weeks) prior to enrollment.
9. Investigational research agents within 28 days (4 weeks) prior to enrollment.
10. Live attenuated vaccines within 28 days (4 weeks) prior to enrollment.
11. Medically indicated subunit or killed vaccines, e.g. influenza, pneumococcal within 2 weeks of initial study vaccine administration unless approved by the study Principal Investigator (PI) or designee
12. Current anti-tuberculosis prophylaxis or therapy.

    -Female-specific criteria:
13. Woman who is breast-feeding or planning to become pregnant during the 24 weeks of study participation.

    -Volunteer has a history of any of the following clinically significant conditions:
14. Serious adverse reactions to vaccines such as anaphylaxis, urticaria (hives), respiratory difficulty, angioedema, or abdominal pain.
15. Clinically significant autoimmune disease or immunodeficiency.
16. Asthma that is not well controlled.
17. Diabetes mellitus (type I or II), with the exception of gestational diabetes.
18. Thyroid disease that is not well controlled.
19. A history of hereditary angioedema (HAE), acquired angioedema (AAE), or idiopathic forms of angioedema.
20. Idiopathic urticaria within the last 1 year.
21. Hypertension that is not well controlled.
22. Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws.
23. Malignancy that is active or history of a malignancy that is likely to recur during the period of the study.
24. Seizure in the past 3 years or treatment for seizure disorder in the past 3 years.
25. Asplenia or functional asplenia.
26. Psychiatric condition that precludes compliance with the protocol; past or present psychoses; or within five years prior to enrollment, history of a suicide plan or attempt.
27. Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer s ability to give informed consent.

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2015-03-26; Primary Completion 2017-04-06 (Actual); Study Completion 2017-04-06 (Actual)

PRIMARY OUTCOMES:
Local and systemic reactogenicity signs and symptoms. | Daily for 7 days following the vaccination
Occurrence of adverse events of all severities. | Through 4 weeks after each injection
Occurrence of serious adverse events and new chronic medical conditions. | Through 48 weeks after last injection

SECONDARY OUTCOMES:
Antibody responses as measured by ELISA and neutralization assays. | 4 weeks after vaccination.
T cell responses as measured by intracellular cytokine staining (ICS)assay. | 4 weeks after vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Julie E Ledgerwood, D.O., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (3):
- United States (3):
  - Hope Clinic - Emory Vaccine Ctr, Decatur, Georgia
  - University of Maryland, Baltimore, Baltimore, Maryland
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland

REFERENCES:
- [Background] Stanley DA, Honko AN, Asiedu C, Trefry JC, Lau-Kilby AW, Johnson JC, Hensley L, Ammendola V, Abbate A, Grazioli F, Foulds KE, Cheng C, Wang L, Donaldson MM, Colloca S, Folgori A, Roederer M, Nabel GJ, Mascola J, Nicosia A, Cortese R, Koup RA, Sullivan NJ. Chimpanzee adenovirus vaccine generates acute and durable protective immunity against ebolavirus challenge. Nat Med. 2014 Oct;20(10):1126-9. doi: 10.1038/nm.3702. Epub 2014 Sep 7. PMID 25194571
- [Background] Ledgerwood JE, DeZure AD, Stanley DA, Coates EE, Novik L, Enama ME, Berkowitz NM, Hu Z, Joshi G, Ploquin A, Sitar S, Gordon IJ, Plummer SA, Holman LA, Hendel CS, Yamshchikov G, Roman F, Nicosia A, Colloca S, Cortese R, Bailer RT, Schwartz RM, Roederer M, Mascola JR, Koup RA, Sullivan NJ, Graham BS; VRC 207 Study Team. Chimpanzee Adenovirus Vector Ebola Vaccine. N Engl J Med. 2017 Mar 9;376(10):928-938. doi: 10.1056/NEJMoa1410863. Epub 2014 Nov 26. PMID 25426834
- [Background] Kibuuka H, Berkowitz NM, Millard M, Enama ME, Tindikahwa A, Sekiziyivu AB, Costner P, Sitar S, Glover D, Hu Z, Joshi G, Stanley D, Kunchai M, Eller LA, Bailer RT, Koup RA, Nabel GJ, Mascola JR, Sullivan NJ, Graham BS, Roederer M, Michael NL, Robb ML, Ledgerwood JE; RV 247 Study Team. Safety and immunogenicity of Ebola virus and Marburg virus glycoprotein DNA vaccines assessed separately and concomitantly in healthy Ugandan adults: a phase 1b, randomised, double-blind, placebo-controlled clinical trial. Lancet. 2015 Apr 18;385(9977):1545-54. doi: 10.1016/S0140-6736(14)62385-0. Epub 2014 Dec 23. PMID 25540891